CLINICAL TRIAL: NCT06302257
Title: Randomized Controlled Trial of Combined Lidocaine - Chlorprocaine in Labor Epidural Analgesia.
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 0532-23-HMO
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Labor Pain
Keywords: Pain; Labor; Analgesia; Local anesthetic; Epidural; Randomized controlled trial; Lidocaine; Chloroprocaine; Visual analogue scale
MeSH Terms: conditions — Labor Pain; Pain; Agnosia | interventions — chloroprocaine; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- lidocaine alone (Active Comparator): Bolus: 20mL MLAC% of lidocaine, administered as incremental test dose over 5 minutes; as in all routine epidurals by our hospital protocol, the incremental test dose is preferred to using classical surgical test doses (which expose the patient to excessive local anesthetic concentrations).
  Interventions: Drug: Lidocaine
- Chlorprocaine only (Experimental): Bolus: 20mL MLAC% of chlorprocaine, administered as incremental test dose over 5 minutes; as above, no other test doses are used.
  Interventions: Drug: Chlorprocaine
- Lidocaine-chlorprocaine combination (Experimental): Bolus: 10mL MLAC% of lidocaine plus 10mL MLAC% of chlorprocaine, mixed in a 20mL syringe, administered as incremental test dose over 5 minutes; as above, no other test doses are used.
  Interventions: Drug: Lidocaine-chlorprocaine combination

INTERVENTIONS:
Drug: Chlorprocaine — we aim to examine whether selective nociceptive analgesia can be obtained in epidural analgesia for women in labor by using a combination of lidocaine (opens TPRV-1 and TPRA-1 channels) and chlorprocaine (polarized local anesthetic)
  Arms: Chlorprocaine only
Drug: Lidocaine — Study participants will receive lidocaine alone
  Arms: lidocaine alone
Drug: Lidocaine-chlorprocaine combination — study participants randomized to this study arm will receive a a 50:50 mixture of both drugs - where all drugs are administered in concentrations based on their ED50 doses, together with epidural opioids (fentanyl)
  Arms: Lidocaine-chlorprocaine combination

SUMMARY:
Abstract: Background: The current "gold standard" epidural analgesia involves some undesirable side effects such as motor and sympathetic blockade. Here, the investigators suggest a new approach for inducing prolonged differential pain blockade during labor by selectively targeting local anesthetic chloroprocaine to the pain-related peripheral (nociceptive) fibers. The investigators approach involves nociceptor-selective anesthesia by selective targeting of ionized local anesthetics into nociceptive fibers via activation of nociceptor-specific TRPV1 channels. The authors demonstrated that activation of these channels by specific TRPV1-agonists (capsaicin or the local anesthetic lidocaine), allows entry of a polarized, membrane-impermeable lidocaine derivative (QX-314) specifically into nociceptive neurons, inhibiting their activity and pain blockade, without causing other neural effects. Capsaicin and QX-314 are not suitable for clinical use, as capsaicin causes severe injection pain and QX-314 is neurotoxic. Here, the investigators use lidocaine as the TRPV1 agonist, and use the high pKa chloroprocaine as the ionized local anesthetic instead of the toxic QX-314. Both drugs are in routine clinical use, but have not been described in co-administration before. The investigators preclinical results show that co-administration of chloroprocaine with TRPV1 agonists, leads to prolonged nociceptor-specific analgesia. KKK Hypothesis: The investigators hypothesize that co-administration of epidural lidocaine (to activate TRPV1 channels) and chloroprocaine (as a polarized local anesthetic which can gain preferential access to nociceptors via opened TRPV1 pores) will elicit selective nociceptive-anesthesia. Methodology: This study assess epidural local analgesia in nulliparous labor. There are 2 stages: Stage 1: Prior to direct comparison of lidocaine (Group L), chloroprocaine (Group C), and a lidocaine-chloroprocaine combination (Group L-C), the investigators first determine equipotential doses of epidural chloroprocaine and lidocaine using double-blinded up-down sequential analysis using the well-established minimum local anesthetic concentration (MLAC or ED50) design. ED50 is estimated using Dixon-Massey analysis and Wilcoxon and Litchfield probit regression. Stage 2: The main phase of the study involves a randomized double-blinded comparison between Groups L, C and L-C where all drug concentrations are based on the ED50/MLAC from the Stage 1. The primary endpoint is a composite measure of selective nociceptive analgesia (VAS pain score / modified Bromage motor score). Secondary outcomes are: 1. pain (VAS 0-100), 2. modified Bromage motor score, 3. thermal imaging of feet and hands, 4. sensory assessment to cold sensation using ice, 5. anesthesia requirement from the PCEA pump, 6. maternal blood pressure. 7. ambulation, and pushing ability in labor. Primary endpoint is assessed using repeated measures ANOVA (first 30-min) and mixed models ANOVA until first analgesic request. Implications: Positive findings will be the first evidence in humans of nociceptor-specific local anesthesia; will provide a more effective neuraxial analgesia protocol for labor, and will lead to future studies of systemic nociceptor-specific local anesthesia.

DETAILED DESCRIPTION:
There are two stages to this study. The first stage requires the determination of equipotential doses of lidocaine and chlorprocaine. The second stage requires randomizing patients to one of three groups - lidocaine alone, chlorprocaine alone, or a mixture of lidocaine and chlorprocaine, in order to assess adequacy of analgesia, the anesthetic dose required, and the presence of non-analgesic effects (such as motor blockade, sensory blockade and sympathetic blockade).

First Stage: Determining equipotential doses of lidocaine and chlorprocaine:

Patients are enrolled early in labor, prior to the request for epidural anesthesia. Epidural analgesia is performed exactly as in routine cases not in the study. Prior to the epidural, patient consent for the epidural is obtained, the patient is placed in the sitting position, the epidural inserted at the L3/4 interspace and a multiport epidural catheter is threaded 3-5 cm into the epidural space. As for routine epidurals in our institution, oxytocin infusions are discontinued during the epidural and are restarted once the patient is comfortable.

Once the epidural is successfully placed (no inadvertent intravascular placement or inadvertent spinal), and if the pre-epidural VAS pain score is >30mm, the patient may be randomized. The patient is assigned to one of the two study drugs (lidocaine or chlorprocaine) using opaque envelopes previously prepared using computer-generated random allocation. As this study is an up-down sequential allocation study, once the drug group is identified, then the specific concentration to be administered is identified from the study log, determined by the success or the failure of the analgesia in the previous patient in the same drug group to the dose of that drug.

Twenty mL cof the study drug is administered as an incremental test dose over the course of 5 minutes. No other test doses are used.

After the final assessment of the study patients are connected to the standard protocol for epidural maintenance and the study is terminated.

Determination of MLAC:As with previous applications of the up-down sequential analysis design in similar studies, the three possible outcomes are "success", "failure" and "reject".

1. Success: Pain during a uterine contraction is measured as either:

   1. VAS ≤ 10mm achieved by 30 minutes from the time of completion of the 20-mL induction dose or b) VAS at least 70 mm less than the VAS immediately prior to the epidural. The consequence of a "success" is that the next patient in that drug group would have a 0.05 % wt/vol reduction in the local anesthetic concentration for the epidural bolus.
2. Failure:Failure is defined as pain during a uterine contraction measured as VAS > 10mm achieved by 30 minutes from the time of completion of the 20mL induction dose, or patient request for supplemental analgesia at that same time point, even if VAS was ≤ 10 mm. The consequence of a "failure" is that the next patient in that drug group would have a 0.05 % wt/vol increase in the local anesthetic concentration for the epidural bolus. The patient will be supplemented with 10 ml (or up to 15 ml if needed) of 1% lidocaine for analgesia.
3. Reject: As for failure (above) but where one of three conditions exist:

   1. rapid progress in labor: repeat vaginal examination at the time of "failure" assessment reveals a cervical dilation of ≥8cm.
   2. top-up doses up to 15 ml of 1 % lidocaine fail to relieve labor pain within a further 20 min (presumably due to failed epidural).
   3. progression to cesarean delivery prior to the 30 min assessment time. The consequence of a "reject" is that the next patient in that group receives the same drug concentration for the epidural bolus.

Measurements The visual analogue pain score (VAPS) is measured during uterine contraction. The anchors for the VAPS are 0 = no pain and 100 = worst pain imaginable.

The following demographic variables are recorded upon enrollment in the study: age, height, weight, gestational age, induction (mode and indication), augmentation, premature rupture of membranes (PROM) and artificial rupture of membranes (AROM). The following obstetric outcome variables are recorded following delivery: 1st stage duration, 2nd stage duration, baby weight, instrumental delivery, Cesarean section for dystocia, Cesarean section for other indications.

The treating anesthesiologist, obstetrician and midwife are blinded to the study group. The patient and all medical personnel, including the anesthesiologist making the assessments, are blinded to the drug group allocation and the drug doses used.

Second phase: The next phase of the study is a randomized controlled study to randomly allocate patients to one of three groups: lidocaine alone, chlorprocaine alone, or a 50:50 mixture of both drugs - where all drugs are administered in concentrations based on their ED50 doses, together with epidural opioids (fentanyl).

Patients are enrolled early in labor, prior to the request for epidural anesthesia. Epidural analgesia is performed exactly as in routine cases not in the study.

Prior to the epidural, patient consent for the epidural is obtained, the VAS pain score is obtained, and the temperature of the feet and hands bilaterally are recorded using a FLIR thermal imaging camera (Flir C3).

The patient is then placed in the sitting position, the epidural inserted at the L3/4 interspace and a multiport epidural catheter is threaded 3-5 cm into the epidural space. As for all routine epidurals in our institution, oxytocin infusions are discontinued during the epidural and are restarted once the patient is comfortable.

As above, once the epidural is successfully placed (no inadvertent intravascular placement or inadvertent spinal), the patient is randomized.

The patient is allocated to one of the three study drug regimes (lidocaine or chlorprocaine or lidocaine-chlorprocaine combination) using opaque envelopes previously prepared using computer-generated random allocation. The concentration to be administered is determined by the ED50 of the previous study (see below).

Three study groups:

Lidocaine only:

Bolus: 20mL MLAC% of lidocaine, administered as incremental test dose over 5 minutes; as in all routine epidurals by our hospital protocol, the incremental test dose is preferred to using classical surgical test doses (which expose the patient to excessive local anesthetic concentrations).

Maintenance: Epidural is connected to a 250mL bag of lidocaine MLAC% + 500mcg fentanyl in 250mL (=2mcg/mL); administered as a PCEA regime with 0 mL/hr background infusion, 10mL bolus dose, 10min lockout time.

Chlorprocaine only:

Bolus: 20mL MLAC% of chlorprocaine, administered as incremental test dose over 5 minutes; as above, no other test doses are used.

Maintenance: Epidural connected to a 250mL bag of lidocaine MLAC% + 500mcg fentanyl in 250mL (=2mcg/mL); administered as PCEA regime with 0 mL/hr background infusion, 10mL bolus dose, 10min lockout time.

Lidocaine-chlorprocaine combination:

Bolus: 10mL MLAC% of lidocaine plus 10mL MLAC% of chlorprocaine, mixed in a 20mL syringe, administered as incremental test dose over 5 minutes; as above, no other test doses are used.

Maintenance: Epidural connected to a 250mL bag containing 125mL lidocaine MLAC% + 125mL chlorprocaine MLAC% + 500mcg fentanyl in 250mL (=2mcg/mL); administered as PCEA regime with 0 mL/hr background infusion, 10mL bolus dose, 10min lockout time.

In keeping with policy for walking epidurals (written protocol from 2005 and recently revived), all patients will be confined to their beds for the first 30 minutes following epidural analgesia and thereafter will be encouraged to ambulate, to go to the bathroom, and to use ambulatory fetal monitors rather than wired fetal monitors. Ambulation, as per our hospital protocol, requires the presence of a member of staff, and the ability to perform knee-bend movements (stand - knee-bend - stand).

Measurements:

The primary endpoint measure at each time point is the composite selective nociceptive analgesia score = VAS pain score / modified Bromage motor block score.

Assessments are made as follows:

1. Pain (VAS 0-100) where the anchors of the VAS score are 0=no pain, 100=worst pain imaginable.

   Need to receive additional anesthesia incase of breakthrough pain and insufficient supplemental doses is also noted.
2. Modified Bromage motor block score where the scores are determined as follows:

1 = unable to move legs or feet; 2 = unable to flex knees, free movement of feet; 3 = just able to flex knees with free movement of feet; 4 = free movement of legs and feet; 5 = able to perform partial knee-bend movements while standing.

3. Thermal imaging of the feet and hands using a FlirC3 thermal camera. Our team have used this technology to identify segmental sympathectomy following spinal anesthesia in mice (Xu Z et al).

4. Sensory assessment to cold sensation using an ice cube (three options - perception of cold, perception of touch, no perception).

5. Anesthesia requirement. From the epidural PCEA pump we will record the frequency of epidural PCA self-administered doses, the need for any rescue supplemental boluses, the numbers of failed attempted self-administered boluses (requests were not allowed because the button was pressed within the 10-minute lockout time), the total dose administered, and the total dose / time of labor.

6. Pushing ability in labor. This will be assessed by the midwife, who is blinded to the study group. As occasionally the delivery of the fetus is impaired by the large size or malrotation of the fetus, this score is assessed not on the successful vaginal delivery, but rather on the strength of pushing and the ability to sense the need to push.

* In the second stage of labor: rate the ability to sense the urge to push: 0-100 (0= complete inability and 100=best imaginable).
* In the second stage of labor: rate the ability push (strength): 0-100 (0= complete inability and 100=best imaginable).

  7. Maternal blood pressure. (Recorded from the fetal heart rate monitor device, as per hospital protocol, every 5 min for the first 20 minutes and every 30 minutes thereafter) Periodicity of assessments VAS pain score is assessed at the peak of uterine contraction. Thermal imaging, cold sensation, and Bromage motor block score are tested (in that order) between uterine contractions. Assessments are made twice at baseline prior to the epidural, and at 10 min intervals for the first 30-minutes, and at 15-minute intervals thereafter until the first epidural top-up request (administered via PCEA).

Anesthesia requirement and pushing ability in labor are recorded at the end of delivery. This includes top up doses (10-15 of Lidocaine 1%) for breakthrough pain.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparity
* Early active labor, cervical dilatation less than 5 cm,
* Age between 18 to 40,
* American Society of Anesthesiologists physical status class II
* Body weight less than 110 kg,
* Gestational age greater than 36 completed weeks,
* Singleton pregnancy
* Vertex presentation.

Exclusion Criteria:

* Narcotic administration in the previous 3 hours
* Previous uterine surgery
* Pre-eclampsia
* Inability to adequately understand the consent

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
VAS pain score / modified Bromage motor block score | 24 Hours
  Pain (VAS 0-100) where the anchors of the VAS score are 0=no pain, 100=worst pain , assesed 30 minutes after placing epidural catheter, , up until the first epidural top-up imaginable.
  Modified Bromage motor block score where the scores are determined as follows:
  1 = unable to move legs or feet; 2 = unable to flex knees, free movement of feet; 3 = just able to flex knees with free movement of feet; 4 = free movement of legs and feet; 5 = able to perform partial knee-bend movements while standing

SECONDARY OUTCOMES:
Segmental sympathectomy | 24 hours
  Thermal imaging of the feet and hands using a FlirC3 thermal camera. Our team have used this technology to identify segmental sympathectomy following spinal anesthesia in mice (Xu Z et al), with use of measuring the temperature of hands and feet
Sensory assessment to cold sensation | 24 hours
  using an ice cube (three options - perception of cold, perception of touch, no perception).For the first 30 minutes after placing the epidural catheter, up until the first epidural top
Anesthesia requirement. | 24 hours
  From the epidural PCEA pump we will record the frequency of epidural PCA self- administered doses, the need for any rescue supplemental boluses, the numbers of failed attempted self-administered boluses (requests were not allowed because the button was pressed within the 10-minute lockout time), the total dose administered, and the total dose / time of labor. For the first 30 minutes after placing the epidural catheter, up until the first epidural top-up
Pushing ability in labor. | 24 hours
  This will be assessed by the midwife, who is blinded to the study group. As occasionally the delivery of the fetus is impaired by the large size or malrotation of the fetus, this score is assessed not on the successful vaginal delivery, but rather on the strength of pushing and the ability to sense the need to push.
  * In the second stage of labor: rate the ability to sense the urge to push: 0-100 (0= complete inability and 100=best imaginable).
  * In the second stage of labor: rate the ability push (strength): 0-100 (0= complete inability and 100=best imaginable). For the first 30 minutes after placing the epidural catheter, up until the first epidural top-up
Maternal Blood pressure | 24 hours
  Assessment will be performed For the first 30 minutes after placing the epidural catheter, up until the first epidural top-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Hebrew University Medical Center, POB 12000, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Undecided